CLINICAL TRIAL: NCT04788446
Title: Develop the Mini-flipped Game-based Learning Strategies in Modified Mediterranean Diet Interventions for Eating Behavior and Cognitive Performance Among Older Adults in the Community
Brief Title: Mediterranean Diet Interventions for Eating Behavior and Cognitive Performance Among Older Adults in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Cheng-Chen Chou, Assistant professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YM109146E
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Healthy
Keywords: Mini-flipped Game-based Learning; Mediterranean Diet; Eating Behavior; Cognitive Performance
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini-flipped Game-based Learning (Experimental): 1. group diet education, an interactive food card game, and guidance on the Mediterranean diet
  2. once a week for 40 minutes.
  3. lasts for 8 weeks
  Interventions: Behavioral: Mini-flipped Game-based Learning
- Balanced diet (Placebo Comparator): 1. given a leaflet on balanced diet and nutrition among the elderly
  2. lasts for 8 weeks
  Interventions: Behavioral: Balanced diet

INTERVENTIONS:
Behavioral: Mini-flipped Game-based Learning — The intervention was 8 weeks, forty minutes adjusted Mediterranean diet learning plan once a week, which includes the 20 minutes for the Mediterranean food table game, and the 20 minutes for the Mediterranean diet nutrition course. The topic of the course includes the relationship between Mediterranean diet and dementia, knowledge of Mediterranean diet, how to integrate local food ingredients into the Mediterranean diet, etc.
  Arms: Mini-flipped Game-based Learning
Behavioral: Balanced diet — Given a balanced diet nutrition health education manual for the aged.
  Arms: Balanced diet

SUMMARY:
The object is to investigate the effects of a modified Mediterranean diet learning intervention program with a Mini-flipped game strategy on dietary behavior and cognitive function of elderly people in the community. The six communities were randomly assigned to the experimental group and the control group. The intervention group will last for 8 weeks. An eight-week Mediterranean diet learning program applying mini-flipped game-based learning strategies could improve dietary behavior and global cognitive function among elderly people living in the general community.

DETAILED DESCRIPTION:
Background：The world is facing an aging population, with an increase in the number of people with mild cognitive impairment and dementia, creating a huge burden of medical costs for individuals, families, and society. Previous studies have shown that the Mediterranean Diet delays cognitive decline, but older adults are less likely to follow the Mediterranean Diet and have less knowledge about the risk of dementia and protective factors of the diet. This study will integrate the Asian version of the Mediterranean Diet Pyramid and local ingredients from Taiwan to design a nutritional health education and game intervention for the Mediterranean Diet.

Purposes：To investigate the effectiveness of developing a Mini-flipped Game-based Learning strategy to promote dietary behavior and cognitive function in the community elderly with a modified diet learning intervention.

Methods：This study was a cluster-randomized controlled trial. The six communities were randomly assigned to the experimental group and the control group.The intervention group completed an eight-week, mini-flipped, game-based learning program reinforcing compliance with the Mediterranean diet, consisting of one 40-minute session per week. The control group members maintained their usual daily diet and were given a booklet on nutrition and health. All participants will be assessed at baseline(0 weeks) and post-test(8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older
* No visual, hearing, or mental impairment, and could speak Mandarin.
* Are willing to participate in the study and fill out the volunteer consent form.

Exclusion Criteria:

* Diagnosis of cognitive dysfunction, brain injury with loss of consciousness for more than 30 minutes, or other central nervous system disorders. The presence of impaired sensory problems.
* Severe illnesses such as heart, liver, and lung failure, end-stage renal disease, total paralysis, terminal cancer or chemotherapy, and a diagnosis of mental illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Mediterranean Diet Score | Change from baseline outcome measure at 8th week (post-test)
  To measure the Mediterranean dietary behavior
Nutrition Knowledge test for the Elderly | Change from baseline outcome measure at 8th week (post-test)
  To measure the nutrition knowledge

SECONDARY OUTCOMES:
Montreal Cognitive Assessment score | Change from baseline outcome measure at 8th week (post-test)
  To measure the objective cognitive function
Cognitive Failures Questionnaire score | Change from baseline outcome measure at 8th week (post-test)
  To measure the subjective cognitive function

OTHER OUTCOMES:
Pittsburgh Sleep Quality Index score | Change from baseline outcome measure at 8th week (post-test)
  To measure the Sleep Quality
Center for Epidemiological Studies Depression Scale score | Change from baseline outcome measure at 8th week (post-test)
  To measure the Depression

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Chen Chou, Principal Investigator — Nursing
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT04788446/Prot_SAP_000.pdf